CLINICAL TRIAL: NCT00474890
Title: A Randomized, Double-Blind, Placebo-Controlled Crossover Study to Assess the Efficacy's Reproducibility of a Combination of Pseudoephedrine and Cetirizine on Symptom Scores and Rhinomanometry in Patients With Allergic Rhinitis Following Pollen Exposure in the Fraunhofer Environmental Challenge Chamber (ECC) in- and Outside the Grass Pollen Season
Brief Title: Study to Compare the Effect of a Combination of Cetirizine With Pseudoephedrine Versus Placebo on Symptoms in Patients With Allergic Rhinitis Within/Out of Season
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 07/03 Inopec ITEM
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Last update posted 2008-02-13 (Estimated); Status verified 2008-02

CONDITIONS: Atopy; Rhinitis
Keywords: Seasonal allergic rhinitis
MeSH Terms: conditions — Rhinitis; Rhinitis, Allergic, Seasonal | interventions — Pseudoephedrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cetericine and pseudoephedrine

SUMMARY:
A previous study has shown very clearly that the treatment with the combination of cetirizine and pseudoephedrine is superior to the treatment with the single agents regarding the reduction of symptoms in patients with allergic rhinitis. These data, obtained after controlled pollen exposure out of the pollen season, showed highly reproducible individual responses prior to dosing. It is not clear, however, whether the same results can be obtained during the pollen season, when additional natural pollen exposure may influence the variability of the individual reactions.

DETAILED DESCRIPTION:
The aim of this study is to evaluate prospectively, if reproducible results can be shown when testing a combination of cetirizine and pseudoephedrine in an Environmental Exposure Unit setting once inside and once outside the grass pollen season. An equivalent outcome would validate the ECC for testing anti-allergic substances during the pollen season in the future. Up to now these studies have been restricted to the pollen-free season.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged 18-55 years. Women will be considered for inclusion if they are:

  * Not pregnant, as confirmed by pregnancy test (see flow chart) and not nursing.
  * Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meet clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit).
  * Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first dose of study medication until at least 72 hours after treatment -, implants, injectables, combined oral contraceptives, some IUDs).
* FEV1 > 80% of predicted at screening.
* Absence of any structural nasal abnormalities or nasal polyps on examination, absence of a history of frequent nose bleeding or recent nasal surgery.
* Absence of conditions or factors, which would make the subject unlikely to be able to stay in the Fraunhofer ECC for 6 hours.
* Non smokers or smokers with a history of less than 10 pack years.
* History of allergic rhinitis to grass pollen and a positive skin prick test for Dactylis glomerata pollen at or within 12 months prior to the screening visit.
* Subject must exhibit a moderate response upon 4000 Dactylis glomerata pollen grains/m3 during 2 hours in the ECC on visit 2
* Subjects with mild stable asthma that is controlled with occasional use of as-needed short-acting beta-agonists and associated with normal lung function may be included.
* Able and willing to give written informed consent to take part in the study.
* Available to complete all study measurements.

Exclusion Criteria:

* Subjects showing clinical symptoms of perennial allergic rhinitis.
* History of a respiratory tract infection and/or exacerbation of asthma within 4 weeks before the screening.
* Any history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnoea, respiratory arrest or hypoxic seizures.
* Administration of oral, injectable or dermal corticosteroids within 8 weeks or intranasal and/or inhaled corticosteroids 4 weeks prior to the screening visit.
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
* Known hypersensitivity, allergic reactions or intolerance to cetirizine, pseudoephedrine or any of the other ingredients.
* Subject receiving monoamine oxidase inhibitors or has received these agents in the last two weeks before dosing.
* Specific Immunotherapy (SIT) within the last two years prior to screening.
* There is a risk of non-compliance with study procedures.
* Participation in another clinical trial 30 days prior to enrolment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2008-02

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Krug, Professor, Principal Investigator — Fraunhofer-Institute of Toxicology and Experimental Medicine
Locations (1):
- Fraunhofer Institute for Toxicology and Experimental Medicine, Hanover, Germany

REFERENCES:
- [Derived] Badorrek P, Dick M, Hecker H, Schaumann F, Sousa AR, Murdoch R, Hohlfeld JM, Krug N. Anti-allergic drug testing in an environmental challenge chamber is suitable both in and out of the relevant pollen season. Ann Allergy Asthma Immunol. 2011 Apr;106(4):336-41. doi: 10.1016/j.anai.2010.12.018. Epub 2011 Feb 5. PMID 21457883